CLINICAL TRIAL: NCT02648490
Title: A Prospective,Open-label, Dose Escalation Phase 1 Study to Investigate the Safety, and Tolerability and to Determine the Maximum Tolerated Dose and Recommended Phase 2 Dose of a HLX07, in Patients With Advanced Solid Cancers.
Brief Title: An Open-label, Phase 1 Study to Determine the Maximum Tolerated Dose of HLX07,in Patients With Advanced Solid Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henlix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX07FIH
Record Dates: First submitted 2015-12-27; First posted 2016-01-07 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2018-03

CONDITIONS: Solid Tumour
Keywords: metastatic or recurrent epithelial cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — HLX07; Acetaminophen; Dexamethasone; Calcium Dobesilate; Diphenhydramine; Ondansetron

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, dose-escalation study of HLX07 ,3+3 design
Oversight: Data Monitoring Committee: No

ARMS (1):
- HLX07, in patients with solid cancers. (Experimental): Each cycle of treatment consists of 4 weeks. Patients who enroll into this study will receive weekly infusion of assigned dose of HLX07. No intra-patient dose escalation is allowed.The proposed dose escalation sequence is 50 mg, 100 mg, 200 mg, 400 mg, 600 mg, 800 mg.
  Acetaminophen 500 mg PO 30 minutes before the infusion of HLX07, followed by dexamethasone 10 mg intravenous infusion for 10 minutes, and followed by diphenhydramine 30 mg intravenous infusion for 10 minutes. If the patient experience grade 2 or 3 nausea and vomiting during the first infusion of HLX07, the addition of 5-HT3 inhibitor may be included in the premedication before subsequent infusions.
  Interventions: Drug: HLX07; Drug: Acetaminophen; Drug: dexamethasone; Drug: diphenhydramine; Drug: 5-HT3 inhibitor

INTERVENTIONS:
Drug: HLX07 — recombinant human anti-EGFR monoclonal antibody against cancers
  Other Names: anti-EGFR monoclonal antibody
Drug: Acetaminophen — Acetaminophen 500 mg PO 30 minutes before the infusion of HLX07.
  Other Names: Tylenol
Drug: dexamethasone — dexamethasone 10 mg intravenous infusion for 10 minutes before the infusion of HLX07.
  Other Names: Decadron; Dexasone
Drug: diphenhydramine — diphenhydramine 30 mg intravenous infusion for 10 minutes before the infusion of HLX07.
  Other Names: Allermax; Benadryl
Drug: 5-HT3 inhibitor — If the patient experience grade 2 or 3 nausea and vomiting during the first infusion of HLX07, the addition of 5-HT3 inhibitor may be included in the premedication before subsequent infusions.
  Other Names: Ondansetron

SUMMARY:
This study is to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of humanized anti-EGFR monoclonal antibody, HLX07, in patients with epithelial cancer who have failed standard therapy and deemed unamenable by conventional therapy. This study will also evaluate the pharmacokinetics, pharmacodynamics, immunogenicity and anti-tumor effect of HLX07 and explore the potential prognostic and predictive biomarkers.

DETAILED DESCRIPTION:
The role of EGFR in carcinogenesis led to the development and extensive evaluation of EGFR-blocking agents for cancer treatment. Two EGFR-targeted approaches have been explored: (a) small-molecule tyrosine kinase inhibitors targeting the intracellular EGFR tyrosine kinase domain and (b). mAbs targeting the EGFR extra-cellular domain.

Small-molecule tyrosine kinase inhibitors have been widely used in lung cancer with EGFR mutations. However, the results of using small molecule inhibitors for cancer with overexpressed wildtype EGFR have been unsatisfactory.

The best-studied of the anti-EGFR mAbs in cancer is cetuximab (Erbitux®), and panitumumab (Vectibix®). Necitumumab, another humanized anti-EGFR mAb is currently under investigation is multiple cancers. Both cetuximab and panitumumab have been approved in colorectal cancer and head/neck cancer.

Cetuximab is chimeric human-murine IgG1 mAb, and blocks ligand binding to EGFR, thereby diminishing receptor dimerization and autophosphorylation and inducing EGFR downregulation. The immunoglobulin IgG1 isotype of cetuximab may also engage hose immune functions such as antibody-dependent cellular cytotoxicity (ADCC). Cetuximab is approved to be used in combination with chemotherapy and has been shown to improve the survival of patients with advanced colorectal cancer. Cetuximab, when used in combination with radiotherapy has also improved response rate in patients with locally advanced head/neck cancer. However, the use of cetuximab has been associated with rare anaphylactic reactions, which is likely to be related to the specific glycosylation in the molecules and possibly its mouse/human chimeric structure.

Panitumumab is a human IgG2 mAb that targets EGFR. But unlike cetuximab, it mediates its effects through mechanisms other than ADCC, which has a different binding site on EGFR extracellular domain from that of cetuximab, is also approved for colorectal cancer and head/neck cancer. However, the side effects, especially skin reactions, is more pronounced in patients receiving panitumumab, which also limiting its clinical use.

Although cetuximab and panitumumab target EGFR, clinical studies of cetuximab and panitumumab have shown that the levels of EGFR expression in cancer cells do not affect the efficacy of the drug.So far there is unclear why it is so. However, several retrospective studies have shown that the presence of K-ras, and B-raf mutations predicts the poor response to either cetuximab or panitumumab. Likewise, there is no clear answer for such phenomenon. Therefore, in this study, the investigators will examine the expression of EGFR in the cancer cells of enrolled patients, but will not use its expression for enrollment. But, in this study, the investigators will exclude patients whose cancer cells harbor either K-ras, or B-raf mutations, since the investigators in vivo study also demonstrated that HLX07 is not effective in cancer cells with K-ras mutations.

HLX07 is an improved version of anti-EGFR monoclonal antibody. There are several important improvements in the development of HLX07. First, the investigators re-engineered the Fab portion of the antibody to modify the glycosylation pattern of this antibody- to make less immunogenic and have better binding affinity. Second, the investigators produced an antibody using CHO cell system, which lead to cleaner glycosylation profile and better yield. Therefore, the investigators expect that the results can provide a better and more affordable option for patients with advanced cancer.

The investigators in vitro and in vivo animal studies have demonstrated that the anti-cancer effect of HLX07 at the same dose level is either equal or superior to those of cetuximab. In the toxicokinetic studies on monkey, the toxicity profile of HLX07 was better than that of cetuximab. Therefore, the investigators are confident that HLX07 will be a better solution for patients who benefit from anti-EGFR monoclonal antibody therapy.

However, HLX07 has not been tested in human yet. Therefore, the investigators propose this first-in-human phase 1 study. In this study, the investigators intend to investigate the safety, and tolerability of HLX07 in humans, and hope to identify the maximum tolerated dose, and determine the recommended phase 2 dose in future study. At the same time, the investigators would like to gain information of the pharmacokinetics and pharmacodynamics of this drug and its potential immunogenicity.

To minimize the risk of patients who volunteer to receive this experimental drug, the investigators will choose 50 mg flat dose as the initial starting dose. The selection of starting dose is based on the repeat-dose toxicology study on monkey. In the 3-month repeat-dose study, the highest non-severely toxic dose (HNSTD) is weekly 60 mg/kg. The human equivalent dose for this HNSTD is 20 mg/kg. One-sixth of 20 mg/kg in an adult of 70 kilogram is 233 mg. In order to provide sufficient safety factor in the FIH study, the investigators will select 50 mg flat dose as the starting dose in this study.

To investigate the dose required to reach maximal effect, the investigators propose a dose escalation sequence. The purpose of the dose escalation is to obtain the pharmacokinetics and pharmacodynamics of HLX07 at different dose levels, and investigate its relationship with adverse reactions. Also, the investigators intend to identify the MTD and determine the dose required to reach 90% saturation of clearance. The information from the dose escalation is crucial to determine the optimal dose in future studies and potential indications for HLX07.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed, unidimensionally-measurable and/or evaluable carcinoma which has failed standard therapy or for whom no standard therapy is available.
2. ECOG performance status score of ≤ 2 at study entry.
3. Able to provide written informed consent.
4. White blood cell (WBC) count ≥3 x 109/L;an absolute neutrophil count ≥ 1.5 x 109/L;a hemoglobin level > 90 g/L; and a platelet count ≥ 100 x 109/L.
5. Adequate hepatic function as defined by: alkaline phosphatase level ≤ 5.0 x the ULN, bilirubin level ≤ 1.5 x the ULN, aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤ 2.5 x the ULN or ≤ 5 x the ULN for patients with liver metastases
6. Adequate renal function as defined by a serum creatinine level within normal limits.
7. Use of effective contraception if procreative potential exists.
8. Life expectancy of approximately 3 months or longer in the opinion of the investigator.

Exclusion Criteria:

1. Chemotherapy, radiation, and/or hormonal therapy (except palliative radiation therapy for disease-related pain and chronic hormonal therapy for prostate carcinoma) within 4 weeks of study entry.
2. Concurrent unstable or uncontrolled medical disease (e.g., active uncontrolled systemic infection, poorly controlled hypertension or history of poor compliance with an anti-hypertensive regimen, unstable angina, congestive heart failure, uncontrolled diabetes) or other chronic disease, which, in the opinion of the investigator, could compromise the patient or the study.
3. Newly-diagnosed or symptomatic brain metastases (patients with a history of brain metastases must have received definitive surgery or radiotherapy, be clinically stable, and not taking steroids; anticonvulsants are allowed).
4. Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. Patients with a previous malignancy but without evidence of disease for more than 3 years will be allowed to enter the trial.
5. Any condition that prevents the patient from providing informed consent.
6. Pregnancy (confirmed by serum beta human chorionic gonadotropin [beta-HCG]) or breast-feeding.
7. Any investigational agent(s) or device(s) within 4 weeks of study entry.
8. Prior treatment with cetuximab, or any other anti-EGFR monoclonal antibody therapy for less than 3 months. Prior treatment with other monoclonal antibodies targeting receptors other than the EGFR is permitted if the drug has been discontinued more than (include) 4 weeks prior to study entry.
9. Tumor cells with either K-ras, N-ras or B-raf mutations.
10. Known history of human immunodeficiency virus infection.
11. Employees of the investigator or study center with direct involvement in this study or other studies under the direction of the investigator or study center, as well as family members of the employees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-09; Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year

SECONDARY OUTCOMES:
Number of participants with treatment-related pathological Complete Response assessed using RECIST 1.1 criteria. | 1 year
  Patients will receive CT/MRI imaging studies every 8 weeks for treatment response until disease progression, withdrawal from the study or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Jiang, Ph.D., Principal Investigator — Henlix, Inc
Locations (2):
- Henlix, Inc., Fremont, California, United States
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hou MM, Ho CL, Lin HY, Zhu Y, Zhang X. Phase I first-in-human study of HLX07, a novel and improved recombinant anti-EGFR humanized monoclonal antibody, in patients with advanced solid cancers. Invest New Drugs. 2021 Oct;39(5):1315-1323. doi: 10.1007/s10637-021-01099-1. Epub 2021 Mar 13. PMID 33713216